CLINICAL TRIAL: NCT00667277
Title: Phase II Study of Bevacizumab (Avastin®) in Myelofibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of response activity in the setting of an unacceptable toxicity profile
Sponsor: Ronald Hoffman (Other)
Collaborators: Myeloproliferative Disorders-Research Consortium (Network); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Ronald Hoffman, Professor of of Medicine, Hematology and Medical Oncology, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 07-0548-00103; P01CA108671-01A2 (NIH); MPD-RC 103 (Other: Myeloproliferative Disorders-Research Consortium)
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Myelofibrosis
Keywords: Myelofibrosis; Idiopathic; Bevacizumab; Avastin; bone marrow fibrosis; bone marrow angiogenesis; JAK2
MeSH Terms: conditions — Primary Myelofibrosis | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bevacizumab (Avastin) (Experimental): Use of bevacizumab (Avastin) in the treatment of myelofibrosis.
  Interventions: Drug: bevacizumab (Avastin)

INTERVENTIONS:
Drug: bevacizumab (Avastin) — 15 mg/kg of bevacizumab by IV infusion once every 3 weeks (1 cycle) for 12 weeks (4 cycles)
  Other Names: Avastin

SUMMARY:
Myelofibrosis is the gradual replacement of bone marrow (place where most new blood cells are produced) by fibrous tissue which reduces the body's ability to produce new blood cells and results in the development of chronic anemia (low red blood cell count). One of the main distinctions of myelofibrosis is "extramedullary hematopoiesis", the migration or traveling of the blood-forming cells out of the bones to other parts of the body, such as the liver or spleen, resulting in an enlarged spleen and liver.

There is not a standard treatment for myelofibrosis, therefore there is no medication that is specifically used in the treatment of myelofibrosis. Bevacizumab (Avastin®) targets and stops a growth factor in the body that helps produce the type of fibrous tissue that is gradually replacing the bone marrow in the bones.

The purpose of this study is to find out how safe and effective bevacizumab is in treating myelofibrosis. The investigators also wish to find out important biologic characteristics or features of myelofibrosis (how it works and operates) during the time of study participation through an additional correlative biomarker study (MPD-RC #107). The purpose of the biomarker study is to understand the causes of MPD and to develop improved methods for the diagnosis and treatment of these diseases, while the main study is trying to find out how well bevacizumab will work in treating the disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary myelofibrosis, essential thrombocythemia related myelofibrosis, and polycythemia vera related myelofibrosis requiring therapy, including those previously treated and relapsed or refractory, or, if newly diagnosed, with intermediate or high risk according to Lille scoring system
* Patients not willing to undergo, not a candidate for, or not having a donor for a bone marrow transplant.
* Signed informed consent: Patients must have signed consents for both the bevacizumab protocol and for the mandatory biomarker MDP-RC 107 protocol to be eligible to participate.
* Patients must have been off any IM-directed therapy for 2 weeks prior to entering this study and have recovered from the toxic effects (grade 0-1) of that therapy.
* Serum bilirubin levels less than or equal to 2 times the upper limit of the normal range for the laboratory (ULN). Higher levels are acceptable if these can be attributed by treating physician to active hemolysis or ineffective erythropoiesis due to myelofibrosis;
* Serum glutamic-pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) levels less than or equal to 2x ULN.
* Serum creatinine levels less than or equal to 1.5 x ULN.
* Women of childbearing potential must have a negative serum or urine pregnancy test prior to bevacizumab treatment and should be advised to avoid becoming pregnant. Men must be advised to not father a child while receiving treatment with bevacizumab. Both women of childbearing potential and men must practice effective methods of contraception (those generally accepted as standard of care measures). Women of child bearing potential are women who are not menopausal for 12 months or who have not undergone previous surgical sterilization.
* Age > 18 years.
* LVEF >50% by MUGA or ECHO (only in patients with prior exposure to anthracyclines).

Exclusion Criteria:

* Nursing and pregnant females. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Inadequately controlled hypertension (defined as systolic blood pressure >140 and/or diastolic blood pressure >90 mmHg on antihypertensive medications) within 4 weeks prior to entering this study
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* Unstable angina
* History of myocardial infarction within 6 months
* History of stroke or transient ischemic attack within 6 months
* History of Budd-Chiari Syndrome or portal vein thrombosis.
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or clinically significant coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days, or anticipation of the need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device or bone marrow biopsy, within 7 days prior to study enrollment
* Proteinuria at screening as demonstrated by either

  * Urine protein:creatinine (UPC) ratio greater than or equal to 1.0 at screening OR
  * Urinalysis with proteinuria ≥ 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).
* History of abdominal fistula, gastrointestinal perforation, peptic ulcer, or intra-abdominal abscess within 6 months
* Ongoing serious, non-healing wound, ulcer, or bone fracture
* Known hypersensitivity to any component of bevacizumab
* Patients with a history of DVT and/or a CNS thrombotic or hemorrhagic event within the past 6 months.
* Patients on anticoagulation therapy for a variety of conditions such as prosthetic heart valves or chronic atrial fibrillation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Hoffman, MD, Principal Investigator — Myeloproliferative Disorders-Research Consortium; Ronald Hoffman, MD, Principal Investigator — Myeloproliferative Disorders Research Consoritum
Locations (5):
- United States (5):
  - Georgetown University, Washington D.C., District of Columbia
  - University of Illinois at Chicago, Chicago, Illinois
  - Weill Cornell, Ithaca, New York
  - Mount Sinai Medical Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Mesa RA, Silver RT, Verstovsek S, Mascarenhas J, Kessler CM, Rondelli D, Goldberg JD, Marchioli R, Demakos EP, Silverman LR, Hoffman R. Single agent bevacizumab for myelofibrosis: results of the Myeloproliferative Disorders Research Consortium Trial. Haematologica. 2013 Sep;98(9):1421-3. doi: 10.3324/haematol.2012.083337. Epub 2013 Jun 28. PMID 23812932

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled in this study between May 2008 and March 2009
Period: Overall Study
Arm/Group | Bevacizumab (Avastin)
Started | 13
Completed | 11
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab (Avastin)
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10
Diagnosis [Number; unit: participants]
  Primary Myelofibrosis (PMF) | 8
  Post-essential Thrombocythemia Myelofibrosis | 3
  Post-Polycythemia Vera Myelofibrosis (Post PV MF) | 2

OUTCOME MEASURES:

1. Primary Outcome: Reason for Therapy Discontinuation
Description: Patient outcomes for myelofibrosis patients treated on a single agent bevacizumab.
  The two subjects who withdrew consent prior to initiation of therapy are included in the "patient refusal" category.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Bevacizumab (Avastin)
Number analyzed (Participants) | 13
participants
  Physician decision | 6
  Patient Refusal | 5
  Death | 1
  End of study | 1

2. Secondary Outcome: Number of Cycles
Description: Number of cycles of bevacizumab received. Patients received bevacizumab as a single agent at a dose of 15 mg/kg intravenously on Day 1 of a 21-day cycle.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: cycles
Arm/Group | Bevacizumab (Avastin)
Number analyzed (Participants) | 11
cycles | 3.1 (2.6)

ADVERSE EVENTS:
Arm/Group | Bevacizumab (Avastin)
Serious Adverse Events (participants affected / at risk) | 7/13
Other Adverse Events (participants affected / at risk) | 7/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (Avastin) (N=13)
Death (Cardiac disorders) | 1 (1) — congestive heart failure
Left Ventricular Failure (Cardiac disorders) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Weight Loss (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (Avastin) (N=13)
Myelo-suppression (Blood and lymphatic system disorders) | 3 (7)
Infection (Skin and subcutaneous tissue disorders) | 1 (1)
Fluid Overload (Vascular disorders) | 1 (1)
General Symptom (General disorders) | 1 (1)
Malaise and Fatigue (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (General disorders) | 1 (1)
Facial Pain (General disorders) | 1 (1)
Bruising (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1)
Infective Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Edema Limbs (Blood and lymphatic system disorders) | 1 (1)
Memory Impairment (Nervous system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Liver Function Test Abnormality (Hepatobiliary disorders) | 1 (4)
Metabolic Laboratory Abnormality (Metabolism and nutrition disorders) | 1 (3)
Protein positive urine (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated due to lack of response activity in the setting of an unacceptable toxicity profile at the completion of the first stage.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes